CLINICAL TRIAL: NCT02525510
Title: A Randomized Trial of Mild Hypothermia and Machine Perfusion in Deceased Organ Donors for Protection Against Delayed Graft Function in Kidney Transplant Recipients
Brief Title: Deceased Organ Donor Interventions to Protect Kidney Graft Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 029669
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Brain Death; Organ Donation; Organ Transplant Failure or Rejection; Delayed Graft Function
Keywords: Mild Hypothermia; Machine Perfusion; Kidney Transplantation
MeSH Terms: conditions — Brain Death; Rejection, Psychology; Delayed Graft Function

STUDY DESIGN:
Intervention Model Description: Enrolled donors will be divided into two populations based on local Organ Procurement Organization criteria:Pump Eligible and Not Pump Eligible.
  Pump Eligible will include three arms. Not Pump Eligible will include two arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Pump Eligible - Normothermia - Pump Both Kidneys (Active Comparator): Normothermia and Machine Perfusion Deceased Donors will be kept normothermic (36.5-37.5 C) prior to organ recovery. Recovered kidneys will receive machine perfusion prior to implantation.
  Interventions: Other: Pump Eligible - Normothermia - Pump Both Kidneys
- Pump Eligible - Hypothermia and Pump Right Kidney (Active Comparator): Deceased Donors will be kept mildly hypothermic (34-35 C) for at least 12 hours prior to organ recovery. Right Kidney will receive machine perfusion prior to implantation and the Left Kidney will receive cold storage.
  Interventions: Other: Pump Eligible - Hypothermia and Pump Right Kidney
- Pump Eligible - Hypothermia and Pump Left Kidney (Active Comparator): Deceased Donors will be kept mildly hypothermic (34-35 C) for at least 12 hours prior to organ recovery. Left Kidney will receive machine perfusion prior to implantation and the Right Kidney will receive cold storage.
  Interventions: Other: Pump Eligible - Hypothermia and Pump Left Kidney
- Not Pump Eligible - Normothermia (Active Comparator): Deceased Donors will be kept normothermic (36.5-37.5 C) prior to organ recovery.
  Interventions: Other: Not Pump Eligible - Normothermia
- Not Pump Eligible - Hypothermia (Active Comparator): Deceased Donors will be kept mildly hypothermic (34-35 C) for at least 12 hours prior to organ recovery.
  Interventions: Other: Not Pump Eligible - Hypothermia

INTERVENTIONS:
Other: Pump Eligible - Normothermia - Pump Both Kidneys — Normothermia and Machine Perfusion Deceased Donors will be kept normothermic (36.5-37.5 C) prior to organ recovery. Recovered kidneys will receive machine perfusion prior to implantation.OPO's protocol
  Arms: Pump Eligible - Normothermia - Pump Both Kidneys
Other: Pump Eligible - Hypothermia and Pump Right Kidney — Deceased Donors will be kept mildly hypothermic (34-35 C) for at least 12 hours prior to organ recovery. Right Kidney will receive machine perfusion prior to implantation and the Left Kidney will receive cold storage.
  Recovered kidneys will be placed in University of Wisconsin for cold storage until reimplantation.
  Arms: Pump Eligible - Hypothermia and Pump Right Kidney
Other: Pump Eligible - Hypothermia and Pump Left Kidney — Deceased Donors will be kept mildly hypothermic (34-35 C) for at least 12 hours prior to organ recovery. Left Kidney will receive machine perfusion prior to implantation and the Right Kidney will receive cold storage.
  Arms: Pump Eligible - Hypothermia and Pump Left Kidney
Other: Not Pump Eligible - Normothermia — Deceased Donors will be kept normothermic (36.5-37.5 C) prior to organ recovery.
  Pulsatile Perfusion of kidney grafts based on the respective OPO's protocol
  Arms: Not Pump Eligible - Normothermia
Other: Not Pump Eligible - Hypothermia — Deceased Donors will be kept mildly hypothermic (34-35 C) for at least 12 hours prior to organ recovery.
  Arms: Not Pump Eligible - Hypothermia

SUMMARY:
To protect kidney function during the transplantation process by comparing mild hypothermia in the deceased organ donor before organs are recovered and pulsatile perfusion of the kidney after recovery and prior to transplantation.

DETAILED DESCRIPTION:
BACKGROUND: In the initial Mild Hypothermia Randomized Control Trial (RCT), in collaboration with the Organ Procurement and Transplant (OPTN) Region 5 Donor Management Goals (DMG) Workgroup and Web Portal, the research team was able to conduct a multi-center RCT examining the benefits of mild hypothermia in donors after neurologic determination of death (DNDDs) on the outcomes of kidney transplantation. The trial was stopped early by the Data and Safety Monitoring Board (DSMB) due to a significant positive benefit to kidney transplant recipients, including a 38% reduction in the odds of delayed graft function (DGF, the primary outcome measure of the trial). The results of this study have been published in the New England Journal of Medicine (July 2015). This research offers a zero-cost intervention that can substantially increase transplant success as well as the pool of potential donors.

To expand upon the success of the hypothermia study, the team is conducting a new RCT to test whether hypothermia is as effective as machine perfusion (MP) of kidneys from DNDDs. In an RCT conducted by the Eurotransplant International Foundation in 2009 (Moers et al. NEJM), the protective effect of MP (OR = 0.57) was similar to that found in the Mild Hypothermia Trial (OR = 0.62). However, the cost of MP can be very significant for organ procurement organizations (OPOs) and transplant centers. MP of kidneys from deceased donors has been increasingly adopted by many centers even though clinical and cost effectiveness studies remain uncertain in the United States. Between 2012 and 2014, out of 31,798 kidneys available for transplant, 11,998 (38%) of them were machine perfused. Over the same three-year period, the number of kidneys pumped annually increased by over 20%. This is an opportune time to investigate the effectiveness of MP compared to mild hypothermia, as there are enough OPOs currently using MP that if mild hypothermia was found to be a non-inferior intervention, there would be considerable cost savings. Similarly, over 60% of kidneys do not receive machine perfusion and findings that demonstrates a benefit of machine perfusion would likely lead to rapid increase in use. In addition, DGF still occurs in up to 56% of high-risk kidneys despite using one of these protective measures and their combined use may be the best approach moving forward. Either way, a new evidence-based standard will be created that will significantly affect the way kidney transplants are handled.

METHODS: This will be a pragmatic multi-site randomized controlled trial that bases enrollment on each OPO/Donation Service Area's current pumping criteria. There will be two main groups of DNDDs,

1. those that are "pump eligible" based on current practice (this group typically resembles traditional expanded criteria donors, but is increased in some areas) and
2. those that are lower risk and whose kidneys do not receive MP ("not pump eligible"). Kidneys from donors who are considered"pump eligible" currently receive MP based on their increased risk for failure. In this trial, "pump eligible" DNDDs will be randomized to one of three groups

(1) normothermia (36.5-37.5 C) plus MP of both kidneys (standard of practice control group), (2) mild hypothermia (34-35 C) plus MP of the left kidney only, and (3) mild hypothermia plus MP of the right kidney only.

In this manner, the same number of kidneys will be randomized to each of the three treatment strategies (MP alone, mild hypothermia alone, or MP + hypothermia). It is important to note that kidneys from "pump eligible"/higher risk DNDDs will still receive one form of protection and possibly two.

In contrast, "not pump eligible" DNDDs will only be randomized to one of two groups: (1) therapeutic mild hypothermia or (2) normothermia. Being that the Mild Hypothermia Trial was stopped early for efficacy in the overall DNDD population, there was insufficient statistical power to confirm a benefit in standard criteria donors (p=0.1 at stoppage). The purpose of this arm of the trial is to validate the protective effect of hypothermia in a larger sample size of lower-risk / "not pump eligible" donors.

The following objectives will be addressed by the trial:

Determine the non-inferiority of a hypothermia-only strategy to a standard pump-only strategy in high risk DNDDs

Evaluate the superiority of a combined hypothermia+MP strategy to both hypothermia or MP alone in high risk DNDDs

Evaluate the superiority of mild hypothermia versus standard of care normothermia in lower risk, "not pump eligible" DNDDs

Determine the safety of the hypothermia strategy with respect to the function of "bystander"organs (e.g., heart, lung)

This protocol has been approved by the OPTN Region 5 Research Committee. In addition, the following steps have been or will be taken:

A National communication was sent via TransplantPro to allow for a two-week period for public comment.

Only donors whose families and/or advanced directives (donor registry) have authorized research will be included in the study.

All organ offers from DNDDs enrolled in the study will include a message in the Donor Highlights section of DonorNet®, a copy of the study summary will be attached to the record, and allocation/transplantation will occur based on standard practice.

There will not be any interaction between the study team and the transplant recipients and no additional data will be collected.

Recipient graft function data will be derived from standard UNet forms and obtained from the OPTN in a de-identified format.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age,
* Brain dead organ donor,
* Authorization for research

Exclusion Criteria:

* Donation after Cardiac Death (DCD) Donor
* Coagulopathy, Hemodynamic instability, Electrolyte deficiencies, Pre-existing kidney disease (per study protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1427 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Delayed Graft Function in Kidney Allografts | 7 days
  The incidence of DGF in kidneys from deceased donors enrolled in this trial, obtained from publically available OPTN data.

SECONDARY OUTCOMES:
Allograft and Recipient survival for all transplanted organs | 1 year
  Allograft and Recipient survival for all transplanted organs from deceased donors enrolled in this trial obtained from publically available OPTN data.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Malinoski, MD, Principal Investigator — Oregon Health and Science University
Locations (7):
- United States (7):
  - Donor Network of Arizona, Phoenix, Arizona
  - U C San Francisco, San Francisco, California
  - Donor Alliance, Denver, Colorado
  - LifeSource, Minneapolis, Minnesota
  - Pacific Northwest Transplant Bank, Portland, Oregon
  - Southwest Transplant Alliance, Dallas, Texas
  - LifeGift, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niemann CU, Feiner J, Swain S, Bunting S, Friedman M, Crutchfield M, Broglio K, Hirose R, Roberts JP, Malinoski D. Therapeutic Hypothermia in Deceased Organ Donors and Kidney-Graft Function. N Engl J Med. 2015 Jul 30;373(5):405-14. doi: 10.1056/NEJMoa1501969. PMID 26222557
- [Background] Jochmans I, Watson CJ. Taking the Heat Out of Organ Donation. N Engl J Med. 2015 Jul 30;373(5):477-8. doi: 10.1056/NEJMe1507573. No abstract available. PMID 26222564
- [Background] Moers C, Smits JM, Maathuis MH, Treckmann J, van Gelder F, Napieralski BP, van Kasterop-Kutz M, van der Heide JJ, Squifflet JP, van Heurn E, Kirste GR, Rahmel A, Leuvenink HG, Paul A, Pirenne J, Ploeg RJ. Machine perfusion or cold storage in deceased-donor kidney transplantation. N Engl J Med. 2009 Jan 1;360(1):7-19. doi: 10.1056/NEJMoa0802289. PMID 19118301
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743
- [Derived] Patel MS, Salcedo-Betancourt JD, Saunders C, Broglio K, Malinoski D, Niemann CU. Therapeutic Hypothermia in Low-Risk Nonpumped Brain-Dead Kidney Donors: A Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2353785. doi: 10.1001/jamanetworkopen.2023.53785. PMID 38416500
- [Derived] Malinoski D, Saunders C, Swain S, Groat T, Wood PR, Reese J, Nelson R, Prinz J, Kishish K, Van De Walker C, Geraghty PJ, Broglio K, Niemann CU. Hypothermia or Machine Perfusion in Kidney Donors. N Engl J Med. 2023 Feb 2;388(5):418-426. doi: 10.1056/NEJMoa2118265. PMID 36724328
- See also: Open Science Framework — https://osf.io/5f3dq/